CLINICAL TRIAL: NCT00987948
Title: Pilot Study of the Effect of Maraviroc Intensification on Peripheral Blood Monocyte HIV DNA Levels When Given to HIV-Infected Subjects Stable on Highly Active Antiretroviral Therapy With Undetectable Plasma HIV RNA
Brief Title: Maraviroc Intensification and Peripheral Blood Monocyte HIV DNA Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H005
Record Dates: First submitted 2009-09-29; First posted 2009-10-01 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: HIV Infections
Keywords: HIV; dementia; High HIV DNA within CD14+ PBMCs; treatment experienced
MeSH Terms: conditions — HIV Infections; Dementia | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Maraviroc (Experimental)
  Interventions: Drug: maraviroc (Selzentry)

INTERVENTIONS:
Drug: maraviroc (Selzentry) — dosage varies with other medications being taken; will follow package insert guidelines

SUMMARY:
High levels of HIV infection within blood monocyte/macrophages (a type of white cells in the bloodstream) increases risk of dementia in HIV-infected individuals. Maraviroc (Selzentry) is a HIV medication that works by blocking the entry of HIV in cells including monocytes/macrophages that use a receptor called CCR5. The study hypothesis is that the addition of Maraviroc to a HIV antiretroviral regimen in HIV-infected individuals with high levels of HIV-infected monocyte/macrophages will lead to a decrease in the levels of infected monocyte/macrophages and to decrease in brain inflammation as studied by magnetic resonance spectroscopy (MRS, a form of MRI study).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection as documented by ELISA and confirmed by either Western blot, HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA by RT-PCR or bDNA at any time prior to study entry.
* Receipt of ARV medication uninterrupted for > 1 year leading up to the screening period with demonstrated HIV RNA < 50 copies/ml for a period of 1 year."
* Willingness for both males and females of childbearing potential to utilize 2 effective contraception methods (2 separate forms, one of which must be an effective barrier method), be non-heterosexually active or have a an exclusive vasectomized partner from screening throughout the duration of the study treatment and for 30 days following the last dose of study drugs.
* Age >18 years.
* Ability and willingness to provide written informed consent
* The following laboratory parameters documented within 30 days prior to study entry:

  * Hemoglobin >8.0
  * Absolute neutrophil count >500
  * Platelet count >40,000
  * AST (SGOT) and ALT (SGPT) <5 x ULN
  * Creatinine <1.5 x ULN
  * Lipase <2.0 x ULN
  * Estimated creatinine clearance > 60 mL/min.
* HIV DNA within peripheral blood mononuclear cells > 100 copies/mL
* Not currently receiving Maraviroc as part of ARV regimen

Exclusion Criteria:

* Past or present HIV opportunistic infection of the brain, learning disability, head injury with prolonged loss of consciousness or cognitive sequelae, or other non-HIV risk factor that may impact cognitive performance.
* Any factor that precludes MRI scan including presence of metal or exposure to metal work (e.g., metal grinder/worker) and claustrophobia
* History of seizure disorder
* History of myocardial infarction, angina, congestive heart failure, peripheral vascular disease, angioplasty or cardiac surgery
* Current malignancy or history of past malignancies excluding basal cell CA
* Any immunomodulator, HIV vaccine, or investigational therapy within 30 days of study entry.
* Any vaccination within 30 days of study entry.
* Requirement for acute therapy for other AIDS-defining illness or other serious medical illnesses (in the opinion of the site investigator) within 14 days prior to study entry.
* Other chronic illnesses including diabetes, autoimmune diseases, and endocrinopathies, except subjects on stable physiologic replacement therapy for low testosterone or thyroid levels
* Known hypersensitivity to Maraviroc
* Any condition which, in the opinion of the investigator, would compromise the subject's ability to participate in the study
* Current active substance or alcohol dependence
* Pregnancy or breast-feeding, intent to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2012-11 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia M Shikuma, M.D., Principal Investigator — University of Hawaii at Manoa
Locations (1):
- Hawaii Center for AIDS, Honolulu, Hawaii, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Maraviroc
Started | 15
Completed | 12
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Maraviroc
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 11
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 24 Weeks in HIV DNA (Log-10 Copies/10^6 Cells) as Measured by HIV DNA Within CD14+ Peripheral Blood Mononuclear Cells
Description: Week 24 minus baseline
Time Frame: Baseline to 24 weeks
Population: Outcome measure in the 12 patients who completed the study.
Measure: Median (Inter-Quartile Range); unit: Log-10 copies/10^6 cells
Arm/Group | Maraviroc
Number analyzed (Participants) | 12
Log-10 copies/10^6 cells | 0.58 [0.00 to 2.20]

2. Secondary Outcome: Change From Baseline to 24 Weeks in Neuropsychological Performance As Measured by Age- and Education-Adjusted Z-Scores
Description: The Z-score represents the number of standard deviations away from the mean, with positive Z-scores representing better neuropsychological performance and negative Z-scores representing poorer neuropsychological performance. Z-scores have been adjusted based on age- and education-matched norms.
Time Frame: Baseline to 24 Weeks
Population: 6 of 12 patients who completed the study who had mild to moderate cognitive impairment
Measure: Median (Inter-Quartile Range); unit: Z-score
Arm/Group | Maraviroc
Number analyzed (Participants) | 6
Z-score | 0.57 [0.35 to 1.07]

ADVERSE EVENTS:
Arm/Group | Maraviroc
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maraviroc (N=15)
Pancreatitis (Endocrine disorders) | 1 (1) — Patient developed abdominal pain at 4 weeks post initiation of study; diagnosed to have pancreatitis. Study medications stopped with resolution of symptoms. SAE assessed as possibly related to maraviroc. MedWatch form filled out.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No